CLINICAL TRIAL: NCT04849949
Title: Acute Consumption of Breakfast Meals With Black Walnut, English Walnuts, or no Nuts
Brief Title: Black Walnuts and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Professor and Director of UGA Obesity Initiative, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AWD00006706
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants in this group received a traditional muffin with butter as the predominant source of fat.
  Interventions: Other: Control
- Black walnut (Experimental): Participants in this group received a muffin in which part of the butter was substituted out for black walnuts.
  Interventions: Other: Black walnut
- English Walnut (Experimental): Participants in this group received a muffin in which part of the butter was substituted out for English walnuts.
  Interventions: Other: English walnut

INTERVENTIONS:
Other: Control — Participants in this group received a traditional muffin with butter as the predominant source of fat.
  Arms: Control
Other: Black walnut — Participants in this group received a muffin in which part of the butter was substituted out for black walnuts.
  Arms: Black walnut
Other: English walnut — Participants in this group received a muffin in which part of the butter was substituted out for English walnuts.
  Arms: English Walnut

SUMMARY:
Walnuts are a nutrient dense food, but most health research is on English walnuts (EW). Black walnuts (BW) contain a different antioxidant and fatty acid profile, and more protein, compared to EW. The purpose of the study was to compare postprandial responses following the consumption of 3 breakfast meals containing either butter (control), BW, or EW.

DETAILED DESCRIPTION:
This study was a randomized, double-blind control trial consisting of 3 study visits for 3 different treatments. The treatments were high-fat breakfast muffins containing either butter (control), black walnuts, or English walnuts. The investigators recruited healthy, normal-weight adults between the ages of 15 and 45y. Study visits were completed in a random order with at least 72 hours between each visit. Anthropometrics, questionnaires, and fasting and postprandial blood samples were collected at each visit.

Hypothesis: The walnut-containing meals would mitigate post-meal increases in glucose, insulin, triglycerides (TG), and lipid peroxidation while improving all measures of subjective appetite and TAC compared to the traditional meal without nuts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women
* Normal-weight (body mass index = 18-24.9kg/m2)

Exclusion Criteria:

* Allergies to test meal ingredients (gluten, eggs, or nuts)
* Medication/supplement usage
* Chronic disease
* Pregnancy or plans to become pregnant
* Special diets
* Tobacco use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Change in triglycerides (TG) and glucose responses | Change from baseline to 3 hours postprandially
  TG (mg/dL) and glucose (mg/dL)
Change in lipid peroxidation | Change from baseline to 3 hours postprandially
  Malondialdehyde (MDA) (uM) measured via Thiobarbituric acid reactive substances (TBARS) assay
Change in total antioxidant capacity | Change from baseline to 3 hours postprandially
  Total antioxidant capacity (uM trolox equivalents) measured via Oxygen Radical Absorbance Capacity (ORAC) assay.
Change in insulin | Change from baseline to 3 hours postprandially
  Insulin (uU/mL)

SECONDARY OUTCOMES:
Change in angiopoietin-like proteins-3 (ANGPTL3) and -4 (ANGPTL4) responses | Change from baseline to 3 hours postprandially
  ANGPTL3 (pg/mL) and ANGPTL4 (pg/mL)
Change in hunger and satiety responses | Change from baseline to 3 hours postprandially
  Hunger, fullness, prospective consumption, and desire to eat measured via a Visual Analog Scale (VAS) (mm). The range of scores on the continuous VAS is 0-100 mm. Zero represents no hunger, fullness, prospective consumption, and desire to eat, while 100 represents the greatest feeling of these outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Paton, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia - Department of Foods and Nutrition & Department of Food Science and Technology, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No